CLINICAL TRIAL: NCT05387096
Title: OPTImization of Medication by Transdisciplinary Assessment of Drug Treatment in Elderly Hospitalized Patients: Application of a Definitive Intervention by Physicians or Clinical Pharmacists
Brief Title: OPTImization of Medication by Transdisciplinary Assessment of Drug Treatment in Elderly Hospitalized Patients
Acronym: OPTIMATE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College Cork (Other)
Collaborators: University Hospital, Ghent (Other); University Hospital Waterford (Other)
Responsible Party: Principal Investigator, Denis O'Mahony, Professor, University College Cork
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DIFA-2020-024
Record Dates: First submitted 2022-04-09; First posted 2022-05-24 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-02

CONDITIONS: Multimorbidity; Polypharmacy
Keywords: inappropriate prescribing; multimorbidity; polypharmacy; hospital admission; older people; frail elderly; medication therapy management; STOPP/START
MeSH Terms: interventions — Potentially Inappropriate Medication List; Pharmacists; methyl 3-mercaptopropionimidate; Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: A randomized controlled clinical trial is proposed in which it is anticipated to randomize 3 x 463 patients to one of 3 groups: (a) standard pharmaceutical care, or (b) trained physician-implemented DI, or (c) clinical pharmacist-implemented DI.
Who Masked: Participant
Masking Description: To mimic the intervention for blinding purposes of the participants, both control and intervention arm patients will receive a sham intervention.While the intervention will be known to clinical staff, the trial statistician will remain blinded until the results are finalized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control: standard pharmaceutical care (Sham Comparator): Patients in the control arm (standard pharmaceutical care) will receive a sham intervention in the form of the modified Medication Adherence Rating Scale (MARS) questionnaire
  Interventions: Other: Sham Intervention
- trained physician-implemented intervention (Active Comparator): The definitive multi-faceted intervention delivered by a trained physician.
  Interventions: Other: Definitive multi-faceted intervention consisting of several components
- clinical pharmacist-implemented intervention (Active Comparator): The definitive multi-faceted intervention delivered by a trained pharmacist.
  Interventions: Other: Definitive multi-faceted intervention consisting of several components

INTERVENTIONS:
Other: Definitive multi-faceted intervention consisting of several components — The definitive intervention will consist of the following components: structured history of medication (SHiM), Screening Tool of Older Persons' Prescriptions (STOPP) and Screening Tool to Alert to Right Treatment (START) screening for PIMs and PPOs, drug-drug and drug-disease interactions screening, face-to-face consultation with attending hospital physicians to discuss PIMs, PPOs, interactions and other issues, pre-discharge medication review and adjustment, detailed medication adjustment discharge report to patients' general practitioners (GPs), post-discharge follow-up contact with patients' GPs and community pharmacists at 1 week, 1 month and 3-6 months post -discharge. The interventions will be applied by a trained physician or pharmacist.
  Other Names: STOPP/START criteria; Face to face consultation with attending physician; medication adjustment report to patient's general practitioner; post discharge follow up with GP and community pharmacist; follow up with patient at 30 and 90-180 days post discharge; the Structured History of Medication (SHiM) questionnaire; Stockley's Drug Interaction Checker
  Arms: clinical pharmacist-implemented intervention; trained physician-implemented intervention
Other: Sham Intervention — Sham intervention in the form of the modified Medication Adherence Rating Scale (MARS) questionnaire in addition to standard care.
  Other Names: Control
  Arms: Control: standard pharmaceutical care

SUMMARY:
This study is being done to find out if a multi-faceted intervention designed to optimize medication in hospitalized older people with multiple chronic medical conditions exposed to multiple medications can reduce unplanned hospital readmission and emergency department attendance compared to current usual medication management. The study intervention aims to minimize potentially inappropriate medications in a structured way and involves follow up with patients and GPs. Patients will be allocated equally to (i) standard medication management (control arm) or (ii) trained physician-delivered intervention or (iii) clinical pharmacist-delivered intervention.

DETAILED DESCRIPTION:
Background:

Recurrent hospitalization and unplanned emergency department (ED) attendance resulting from potentially inappropriate medication is an increasingly common phenomenon in older people with multi-morbidity and associated polypharmacy. With a growing older population with multi-morbidity/polypharmacy, there is a pressing need to address the increasing challenge of potentially inappropriate medications (PIMs) and potential prescribing omissions (PPOs) and associated problems that accentuate adverse drug reactions/events and avoidable excess morbidity. There is also an imperative to curb excess healthcare expenditure related to preventable medication-related problems.

Objective:

To test the clinical and economic impact of a multi-faceted medication optimization definitive intervention on avoidable rehospitalization and unscheduled ED attendance in multi-morbid patients aged ≥ 70 years hospitalized with acute illness.To test the clinical and economic impact of a multi-faceted medication optimization definitive intervention (DI) on avoidable rehospitalization and unscheduled ED attendance in multi-morbid patients aged ≥ 70 years hospitalized with acute illness.

Design:

A randomized controlled clinical trial is proposed in which it is anticipated to randomize 3 x 463 patients to one of 3 groups: (a) standard pharmaceutical care, or (b) trained physician-implemented DI, or (c) clinical pharmacist-implemented DI.

Setting: Acute care environment in 3 large tertiary referral teaching hospitals with similar custom and practice relating to management of older people with acute illness.

Participants: Patients aged ≥ 70 years with multi-morbid illness i.e. ≥ 3 chronic medical conditions and associated polypharmacy i.e. ≥ 5 daily prescription medications admitted with acute unselected illness.

Intervention:

The definitive multi-faceted intervention will consist of the following components:modified structured history of medication (SHiM), Screening Tool of Older Persons' Prescriptions (STOPP) and Screening Tool to Alert to Right Treatment (START) screening for PIMs and PPOs using STOPP/START version 3.0, drug-drug interaction screening using Stockley's Drug Interaction Checker, face-to-face consultation with attending hospital physicians to discuss PIMs, PPOs, interactions and other issues, pre-discharge medication review and adjustment, detailed medication adjustment discharge report to patients' general practitioners (GPs), post-discharge follow-up contact with patients' GPs and community pharmacists at 1 week and 1 and 3-6 months post-discharge.

Study Population:

OPTIMATE will focus on patients admitted with acute medical or surgical illness to Cork University Hospital, University Hospital Waterford and Ghent University Hospital. Patients to be screened for enrolment are those admitted primarily under the care of specialist departments other than geriatric medicine.

Data Collection:

All OPTIMATE trial data will be collected electronically and entered on a bespoke trial proforma. Once verified as fully correct and complete, all individual participant trial data will be stored on a fully secure clinical trial database.

Statistical Analysis:

Treatment effects for each of the two active intervention arms (versus control) in terms of binary outcomes (e.g. readmission) will be estimated using logistic regression, while Health Related QoL (EQ-5D 5L) will be analyzed using ordinal regression with a logit link function (i.e. a proportional odds model). We will report two models for each outcome: one adjusted for centre and admitting service type; and another further adjusted for centre, age (years), sex, number of comorbidities at baseline, and number of prescribed medications at baseline. Effect estimates will be reported as odds-ratios with 95% confidence intervals and exact p-values. There will be no correction for multiplicity, but we will report results for all outcomes regardless of the result and provide enough information for the reader to make whatever corrections they may consider appropriate. Equivalence tests comparing the two active arms (for each outcome) will be done using a "two one-sided tests" procedure based on a 90% confidence interval (which equates to a 5% type 1 error rate). All analyses will be conducted on an intention-to-treat basis and will be conducted under the quality system and SOPs of the HRB CRF-C Statistics and Data Analysis Unit. A complete statistical analysis plan (SAP) will be pre-registered on the Open Science Framework prior to patient recruitment database lock. Any necessary deviations from this SAP will be documented and explained in the trial report. There will be only one single trial data analysis at the end of the project. All reporting will be carried out in accordance with CONSORT guidelines for clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 70years
2. 3 or more chronic conditions.
3. ≥ 5 daily medications pre-admission, all medications taken for at least 4 weeks continuously.
4. Can speak and understand English (in the two Irish medical centres), and Dutch or French in Ghent University Hospital (Ghent is predominantly Dutch-speaking).
5. Can give informed consent or give witnessed verbal consent or have a suitable proxy who can give informed assent on the patient's behalf.
6. Agrees to follow-up contact post-discharge up to 180 days post-randomization.
7. Agrees to primary researcher contacting the GP and community pharmacist post-discharge.

Exclusion Criteria:

1. Terminal illness.
2. Severe dementia and clearly unable to understand the purpose of the trial or give consent to participation.
3. Severe communication disorder, making informed consent impossible.
4. Likely to be discharged from hospital within 48 hours of arrival.
5. Intensive Care Unit (ICU) admission.
6. Primary psychiatric presenting illness.
7. Unavailable for post-discharge follow-up for any reason.
8. Non-accidental poisoning.
9. Previous participation in medication optimization trials.
10. Active participation in another clinical trial
11. Infectious illness requiring strict isolation (including COVID-19 infection) blocking access of the primary researcher to the patient for enrolment.
12. End-stage renal, liver or lung disease requiring organ replacement therapy.
13. Admitted under the care of specialists in Clinical Pharmacology, Palliative Medicine, Clinical Oncology or Haematology.
14. Admitted under the care of specialists in Geriatric Medicine in Ghent University Hospital.
15. Trial participation refusal.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 642 (Actual)
Dates: Start 2023-01-17 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Unscheduled readmission to hospital. | At day 30 post-discharge.
  All-cause re-hospitalization in multi-morbid older people exposed to polypharmacy. Computerized hospital admission records will be inspected. If hospital readmission has occurred dates of admission and discharge will be recorded in the electronic case report form.
Emergency Department attendance. | At day 30 post-discharge.
  Unscheduled emergency department attendance at in multi-morbid older people exposed to polypharmacy. Computerized hospital emergency department attendance records will be inspected. The primary researcher will record on the electronic case report form whether there has there been an unscheduled emergency department attendance since the first follow-up post discharge.
Composite endpoint 1 | At day 30 post-discharge.
  Composite endpoint of readmission to hospital or emergency department attendance within 30 days of discharge from the index admission.
Unscheduled readmission to hospital. | At between days 90 and 180 post-discharge.
  Unscheduled readmission at 180 days post-discharge in multi-morbid older people exposed to polypharmacy. This will be ascertained during the follow-up interview within 180 (+/-14) days post-discharge. Computerized hospital emergency department attendance records will be inspected. The primary researcher will record on the electronic case report form whether there has there been an unscheduled readmission at 180 days since discharge from the index hospital admission.
Emergency Department attendance. | At between days 90 and 180 post-discharge.
  Unscheduled emergency department attendance at in multi-morbid older people exposed to polypharmacy. This will be ascertained during the follow-up interview within 180 (+/-14) days post-discharge. Computerized hospital emergency department attendance records will be inspected. The primary researcher will record on the electronic case report form whether there has there been an unscheduled emergency department attendance at 180 days since discharge from the index hospital admission.
Composite endpoint 2 | At between days 90 and 180 post-discharge.
  Composite endpoint of readmission to hospital or emergency department attendance within 180 days of discharge from the index admission.

SECONDARY OUTCOMES:
Quality of life measured by EuroQol quality of life 5 dimensional 5 level instrument (incorporating pain control) | At day 30 post-discharge.
  The EuroQol quality of life 5 dimensional 5 level instrument (EQ5D-5L) is a self-reported quality of life questionnaire comprised of five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each of the five dimensions is divided into five levels: level 1 (no problem), level 2 (slight problems), level 3 (moderate problems), level 4 (severe problems) and level 5 (unable to/extreme problems).The results are used to calculate a five digit score that describes the patient's health state. This value is the converted into an index value, on a range between 0 and 1, where 0 represents "a state as bad as being dead" and 1 represents "full health".In addition, the questionnaire has a Visual Analogue Scale question which asks the patient to indicate their overall health on the day of questionnaire completion. This is a 0 -100 scale where 100 represents "The best health you can imagine' and 0 'The worst health you can imagine'.
Quality of life measured by EuroQol quality of life 5 dimensional 5 level instrument | At between days 90 and 180 post-discharge.
  The EQ5D-5L is a self-reported quality of life questionnaire comprised of five dimensions. The questionnaire gives a score in the range between 0 and 1, where 0 represents "a state as bad as being dead" and 1 represents "full health".In addition, the questionnaire has a Visual Analogue Scale question which asks the patient to indicate their overall health on the day of questionnaire completion. This is a 0 -100 scale where 100 represents "The best health you can imagine' and 0 'The worst health you can imagine'.
All-cause mortality | At day 30 post-discharge.
  secondary outcome
All-cause mortality | At between days 90 and 180 post-discharge.
  secondary outcome
Occurrence of first admission to residential care facility for long-term nursing care | At day 30 post-discharge.
  secondary outcome
Occurrence of first admission to residential care facility for long-term nursing care | At between days 90 and 180 post-discharge.
  secondary outcome

OTHER OUTCOMES:
Quality Life Adjusted Year (QALY) | At between days 90 and 180 post-discharge.
  The study proposes to examine the DI cost-effectiveness from the wider public health services perspective including possible costs and benefits accrued via the community services and rehospitalizations. The study aims to assess the following cost-effectiveness measures of the DI as delivered by a trained physician and by a trained pharmacist
Cost per hospital readmission avoided | At between days 90 and 180 post-discharge.
  The cost-effectiveness analysis will be performed by combining quality of life data and data from hospital records (the number of days in hospital if readmitted) and health resource utilization costs.
Cost per ED attendance avoided | At between days 90 and 180 post-discharge.
  The cost-effectiveness analysis will be performed by combining quality of life data and data from hospital records (the number of emergency department attendances and health resource utilization costs.
Unscheduled readmission to hospital within 180 days of discharge | At between days 90 and 180 post-discharge.
  All-cause re-hospitalization in multi-morbid older people exposed to polypharmacy. This will be ascertained during the follow-up interview within 180 (+/-14) days post-discharge. The primary researcher will record on the electronic case report form whether there has there been an unscheduled hospital admission. Computerized hospital admission records will be inspected. If hospital readmission has occurred dates of admission and discharge will be recorded in the electronic case report form.
Composite endpoint of readmission to hospital or emergency department attendance within 180 days of discharge | At between days 90 and 180 post-discharge.
  All-cause re-hospitalization (outcome 2) will be ascertained as described. The number of days in hospital will be calculated for each visit and from these figures, the total days in hospital will be calculated. Unscheduled emergency department attendance (outcome 3) will also be ascertained as described. Computerized admission and emergency department attendance records will be used. The composite endpoint will be calculated from outcomes 2 and 3.

CONTACTS AND LOCATIONS:
Overall Officials: Denis O'Mahony, Professor, Principal Investigator — University College Cork
Locations (3):
- Ghent University Hospital, Ghent, Belgium
- Ireland (2):
  - Cork University Hospital, Cork
  - University Hospital Waterford, Waterford

IPD SHARING:
Plan to Share IPD: Yes
Consent from patients participating in OPTIMATE will be obtained for all data to be shared publicly, such as data used in the generation of publications arising from the study. Data sharing repositories will be formerly identified via careful alignment of the expected data object outputs and evaluated using the re3data resource (re3data.org). This is to ensure maximum utility and interoperability of the final data package(s) and assignment of a persistent digital object identifier (DOI). Additional post-study data provenance will be enacted through sharing of analysis scripts and study protocols via Open Science Framework projects with an accompanying DOI(s) and/or through the Health Research Board (HRB) Open Research publishing platform.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be made available six months after publication.
Access Criteria: Open access

REFERENCES:
- [Background] Al Hamid A, Ghaleb M, Aljadhey H, Aslanpour Z. A systematic review of hospitalization resulting from medicine-related problems in adult patients. Br J Clin Pharmacol. 2014 Aug;78(2):202-17. doi: 10.1111/bcp.12293. PMID 24283967
- [Background] Blum MR, Sallevelt BTGM, Spinewine A, O'Mahony D, Moutzouri E, Feller M, Baumgartner C, Roumet M, Jungo KT, Schwab N, Bretagne L, Beglinger S, Aubert CE, Wilting I, Thevelin S, Murphy K, Huibers CJA, Drenth-van Maanen AC, Boland B, Crowley E, Eichenberger A, Meulendijk M, Jennings E, Adam L, Roos MJ, Gleeson L, Shen Z, Marien S, Meinders AJ, Baretella O, Netzer S, de Montmollin M, Fournier A, Mouzon A, O'Mahony C, Aujesky D, Mavridis D, Byrne S, Jansen PAF, Schwenkglenks M, Spruit M, Dalleur O, Knol W, Trelle S, Rodondi N. Optimizing Therapy to Prevent Avoidable Hospital Admissions in Multimorbid Older Adults (OPERAM): cluster randomised controlled trial. BMJ. 2021 Jul 13;374:n1585. doi: 10.1136/bmj.n1585. PMID 34257088
- [Background] Cardwell K. Reducing medication errors and transitions of care. Age Ageing. 2020 Jul 1;49(4):537-539. doi: 10.1093/ageing/afaa065. No abstract available. PMID 32474582
- [Background] Dalton K, O'Mahony D, O'Sullivan D, O'Connor MN, Byrne S. Prescriber Implementation of STOPP/START Recommendations for Hospitalised Older Adults: A Comparison of a Pharmacist Approach and a Physician Approach. Drugs Aging. 2019 Mar;36(3):279-288. doi: 10.1007/s40266-018-0627-2. PMID 30659429
- [Background] Drenth-van Maanen AC, Spee J, van Hensbergen L, Jansen PA, Egberts TC, van Marum RJ. Structured history taking of medication use reveals iatrogenic harm due to discrepancies in medication histories in hospital and pharmacy records. J Am Geriatr Soc. 2011 Oct;59(10):1976-7. doi: 10.1111/j.1532-5415.2011.03610_11.x. No abstract available. PMID 22091519
- [Background] El Morabet N, Uitvlugt EB, van den Bemt BJF, van den Bemt PMLA, Janssen MJA, Karapinar-Carkit F. Prevalence and Preventability of Drug-Related Hospital Readmissions: A Systematic Review. J Am Geriatr Soc. 2018 Mar;66(3):602-608. doi: 10.1111/jgs.15244. Epub 2018 Feb 22. PMID 29468640
- [Background] Hyttinen V, Jyrkka J, Valtonen H. A Systematic Review of the Impact of Potentially Inappropriate Medication on Health Care Utilization and Costs Among Older Adults. Med Care. 2016 Oct;54(10):950-64. doi: 10.1097/MLR.0000000000000587. PMID 27367864
- [Background] Kongkaew C, Noyce PR, Ashcroft DM. Hospital admissions associated with adverse drug reactions: a systematic review of prospective observational studies. Ann Pharmacother. 2008 Jul;42(7):1017-25. doi: 10.1345/aph.1L037. Epub 2008 Jul 1. PMID 18594048
- [Background] Kuhn-Thiel AM, Weiss C, Wehling M; FORTA authors/expert panel members. Consensus validation of the FORTA (Fit fOR The Aged) List: a clinical tool for increasing the appropriateness of pharmacotherapy in the elderly. Drugs Aging. 2014 Feb;31(2):131-40. doi: 10.1007/s40266-013-0146-0. PMID 24353033
- [Background] Laugaland K, Aase K, Barach P. Interventions to improve patient safety in transitional care--a review of the evidence. Work. 2012;41 Suppl 1:2915-24. doi: 10.3233/WOR-2012-0544-2915. PMID 22317162
- [Background] Lavan A, Eustace J, Dahly D, Flanagan E, Gallagher P, Cullinane S, Petrovic M, Perehudoff K, Gudmondsson A, Samuelsson O, Sverrisdottir A, Cherubin A, Dimitri F, Rimland J, Cruz-Jentoft A, Velez-Diaz-Pallares M, Lozano Montoya I, Soiza RL, Subbarayan S, O'Mahony D. Incident adverse drug reactions in geriatric inpatients: a multicentred observational study. Ther Adv Drug Saf. 2018 Jan;9(1):13-23. doi: 10.1177/2042098617736191. Epub 2017 Oct 24. PMID 29318003
- [Background] Leendertse AJ, Van Den Bemt PM, Poolman JB, Stoker LJ, Egberts AC, Postma MJ. Preventable hospital admissions related to medication (HARM): cost analysis of the HARM study. Value Health. 2011 Jan;14(1):34-40. doi: 10.1016/j.jval.2010.10.024. PMID 21211484
- [Background] McAuliffe LH, Zullo AR, Dapaah-Afriyie R, Berard-Collins C. Development and validation of a transitions-of-care pharmacist tool to predict potentially avoidable 30-day readmissions. Am J Health Syst Pharm. 2018 Feb 1;75(3):111-119. doi: 10.2146/ajhp170184. PMID 29371191
- [Background] Moriarty F, Bennett K, Cahir C, Kenny RA, Fahey T. Potentially inappropriate prescribing according to STOPP and START and adverse outcomes in community-dwelling older people: a prospective cohort study. Br J Clin Pharmacol. 2016 Sep;82(3):849-57. doi: 10.1111/bcp.12995. Epub 2016 Jun 9. PMID 27136457
- [Background] O'Brien GL, O'Mahony D, Gillespie P, Mulcahy M, Walshe V, O'Connor MN, O'Sullivan D, Gallagher J, Byrne S. Cost-Effectiveness Analysis of a Physician-Implemented Medication Screening Tool in Older Hospitalised Patients in Ireland. Drugs Aging. 2018 Aug;35(8):751-762. doi: 10.1007/s40266-018-0564-0. PMID 30003429
- [Background] O'Connor MN, O'Sullivan D, Gallagher PF, Eustace J, Byrne S, O'Mahony D. Prevention of Hospital-Acquired Adverse Drug Reactions in Older People Using Screening Tool of Older Persons' Prescriptions and Screening Tool to Alert to Right Treatment Criteria: A Cluster Randomized Controlled Trial. J Am Geriatr Soc. 2016 Aug;64(8):1558-66. doi: 10.1111/jgs.14312. Epub 2016 Jul 1. PMID 27365262
- [Background] O'Mahony D, O'Sullivan D, Byrne S, O'Connor MN, Ryan C, Gallagher P. STOPP/START criteria for potentially inappropriate prescribing in older people: version 2. Age Ageing. 2015 Mar;44(2):213-8. doi: 10.1093/ageing/afu145. Epub 2014 Oct 16. PMID 25324330
- [Background] O'Mahony D, Gudmundsson A, Soiza RL, Petrovic M, Cruz-Jentoft AJ, Cherubini A, Fordham R, Byrne S, Dahly D, Gallagher P, Lavan A, Curtin D, Dalton K, Cullinan S, Flanagan E, Shiely F, Samuelsson O, Sverrisdottir A, Subbarayan S, Vandaele L, Meireson E, Montero-Errasquin B, Rexach-Cano A, Correa Perez A, Lozano-Montoya I, Velez-Diaz-Pallares M, Cerenzia A, Corradi S, Soledad Cotorruelo Ferreiro M, Dimitri F, Marinelli P, Martelli G, Fong Soe Khioe R, Eustace J. Prevention of adverse drug reactions in hospitalized older patients with multi-morbidity and polypharmacy: the SENATOR* randomized controlled clinical trial. Age Ageing. 2020 Jul 1;49(4):605-614. doi: 10.1093/ageing/afaa072. PMID 32484850
- [Background] O'Sullivan D, O'Mahony D, O'Connor MN, Gallagher P, Gallagher J, Cullinan S, O'Sullivan R, Eustace J, Byrne S. Prevention of Adverse Drug Reactions in Hospitalised Older Patients Using a Software-Supported Structured Pharmacist Intervention: A Cluster Randomised Controlled Trial. Drugs Aging. 2016 Jan;33(1):63-73. doi: 10.1007/s40266-015-0329-y. PMID 26597401
- [Background] Oscanoa TJ, Lizaraso F, Carvajal A. Hospital admissions due to adverse drug reactions in the elderly. A meta-analysis. Eur J Clin Pharmacol. 2017 Jun;73(6):759-770. doi: 10.1007/s00228-017-2225-3. Epub 2017 Mar 1. PMID 28251277
- [Background] Ravn-Nielsen LV, Duckert ML, Lund ML, Henriksen JP, Nielsen ML, Eriksen CS, Buck TC, Pottegard A, Hansen MR, Hallas J. Effect of an In-Hospital Multifaceted Clinical Pharmacist Intervention on the Risk of Readmission: A Randomized Clinical Trial. JAMA Intern Med. 2018 Mar 1;178(3):375-382. doi: 10.1001/jamainternmed.2017.8274. PMID 29379953
- [Background] Thomsen LA, Winterstein AG, Sondergaard B, Haugbolle LS, Melander A. Systematic review of the incidence and characteristics of preventable adverse drug events in ambulatory care. Ann Pharmacother. 2007 Sep;41(9):1411-26. doi: 10.1345/aph.1H658. Epub 2007 Jul 31. PMID 17666582
- [Background] Thompson K, Kulkarni J, Sergejew AA. Reliability and validity of a new Medication Adherence Rating Scale (MARS) for the psychoses. Schizophr Res. 2000 May 5;42(3):241-7. doi: 10.1016/s0920-9964(99)00130-9. PMID 10785582
- [Background] Weir DL, Lee TC, McDonald EG, Motulsky A, Abrahamowicz M, Morgan S, Buckeridge D, Tamblyn R. Both New and Chronic Potentially Inappropriate Medications Continued at Hospital Discharge Are Associated With Increased Risk of Adverse Events. J Am Geriatr Soc. 2020 Jun;68(6):1184-1192. doi: 10.1111/jgs.16413. Epub 2020 Mar 31. PMID 32232988
- [Background] Xing XX, Zhu C, Liang HY, Wang K, Chu YQ, Zhao LB, Jiang C, Wang YQ, Yan SY. Associations Between Potentially Inappropriate Medications and Adverse Health Outcomes in the Elderly: A Systematic Review and Meta-analysis. Ann Pharmacother. 2019 Oct;53(10):1005-1019. doi: 10.1177/1060028019853069. Epub 2019 May 25. PMID 31129978
- [Background] Cullinan S, O'Mahony D, Byrne S. Application of the structured history taking of medication use tool to optimise prescribing for older patients and reduce adverse events. Int J Clin Pharm. 2016 Apr;38(2):374-9. doi: 10.1007/s11096-016-0254-0. Epub 2016 Jan 21. PMID 26797770
- See also: Drug-drug interaction tool — https://www.pharmaceuticalpress.com/products/stockleys-drug-interactions/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-13): https://cdn.clinicaltrials.gov/large-docs/96/NCT05387096/Prot_SAP_000.pdf